CLINICAL TRIAL: NCT04744727
Title: Efficacy and Safety of Intravenous Paracetamol in Manament of Labour Pain in a Low Resource Setting
Brief Title: Efficacy and Safety of Intravenous Paracetamol in Manament of Labour Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, lecturer of obstetrics and gynecology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/2019OBSGN/27
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Cases were divided into 2 groups:
  Group I (paracetamol group): Included 48 pregnant women who received 1000 mg of intravenous paracetamol. The treatment was administered at the begining of the active phase of 1st stage of labor [roughly defined as a cervical dilatation of 3-4 cm and a cervical effacement ≥ 50%].
  Group 2 (pethidine group): Included 48 pregnant women who received 50 mg of intravenous pethidine HCL diluted in 10 ml normal saline. The treatment was administered at the beginning of the active phase of 1st stage of labor [roughly defined as a cervical dilatation of 3-4 cm and a cervical effacement ≥ 50%]. Randomization was done by a computer-generated randomization system. Letters of the allocated were concealed in serially numbered opaque envelope that were only released after recruitment.
Who Masked: Participant
Masking Description: Letters of the allocated were concealed in serially numbered opaque envelope that were only released after recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paracetamol group (Active Comparator): Included 48 pregnant women who received 1000 mg of intravenous paracetamol. The treatment was administered at the begining of the active phase of 1st stage of labor [roughly defined as a cervical dilatation of 3-4 cm and a cervical effacement ≥ 50%].
  Interventions: Drug: paracetamol-pethidine
- pethidine group (Active Comparator): Included 48 pregnant women who received 50 mg of intravenous pethidine HCL diluted in 10 ml normal saline. The treatment was administered at the beginning of the active phase of 1st stage of labor [roughly defined as a cervical dilatation of 3-4 cm and a cervical effacement ≥ 50%].
  Interventions: Drug: paracetamol-pethidine

INTERVENTIONS:
Drug: paracetamol-pethidine — 100 ml containing 1000 mg paracetamol -50 mg pethidine HCL

SUMMARY:
to compare between the use of single dose of paracetamol and pethidine hydrochloride intravenously in management of labour pains

DETAILED DESCRIPTION:
investigators conducted a randomized clinical study included including 96 primiparous women admitted to Obstetrics and Gynecology Department, Menoufia University Hospitals, starting the study from May 2019 to March 2020 to assess the use of paracetamol intravenously versus Pethidine HCL intravenously in management of intrapartum pain. After obtaining approval from the local ethics committee, women who agreed to participate gave their signed informed consent after explanation of the trial benefits and hazards

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* aged 18-35 years,
* Term live singleton pregnancy,
* Vertex presentation,
* Spontaneous onset of labor at term 37-42 weeks gestation,
* In active phase of of 1st stage of labour (cervix dilatation 3- 4 cm).

Exclusion Criteria:

Clinical evidence of cephalopelvic disproportion

* Use of any kind of analgesia prior to study
* Any medical disorder during pregnancy (liver or kidney impairment)
* Induction of labor, Intrauterine fetal death
* Evidence of fetal distress
* Antenatal diagnosis of congenital malformation
* Previous history of hypersensitivity to either drug
* Extremes of age (i.e. below 18 or above 35)
* Multiple pregnancies
* Cervical dilatation more than 6 cm.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
change of the intensity of perceived labor pain. | immediately after the intervention and up to 3 hours after the intervension
  Labour pain was semi-objectively assessed using the visual analogue scale (VAS). In this technique, the patient is shown a ten cm line which represent at one end no pain and the other worst pain, and the patient is asked to point on the line where her pain lies. This scale has the added advantage that the pain can be given a numerical value.

SECONDARY OUTCOMES:
duration of the active phase of the 1st stage of labor | immediately from start of active phase of the 1st stage of labor till the end of first stage
duration of the 2nd stage of labor | immediately from start of second stage till deliver of fetus
need for further analgesia | immediately after the intervention till the end of first stage of labour
maternal dizziness, nausea and/or vomiting | immediately after the intervention till the end of first stage
mode of delivery (vaginal or by caesarian | immediately after the intervention
1- and 5-minutes Apgar scores. | immediately after delivery of the fetus
need for neonatal resuscitation | immediately after delivery of the fetus
need for NICU admission | immediately after delivery of the fetus
Neonatal respiratory distress . | immediately after delivery of the fetus

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Anter, Study Director — Faculty of medicine-Menoufia university-shebin elkom -egypt
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

REFERENCES:
- [Derived] Anter ME, Abdel Attey Saleh S, Shawkey Allam S, Mohamed Nofal A. Efficacy and safety of intravenous paracetamol in management of labour pains in a low resource setting: a randomized clinical trial. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6320-6328. doi: 10.1080/14767058.2021.1911995. Epub 2021 Apr 26. PMID 33902372